CLINICAL TRIAL: NCT03897790
Title: Evaluation of Transcranial Doppler Vasoconstrictor Vasoreactivity During General Anesthesia in Hypertensive Patients
Acronym: DiVADH
Status: Withdrawn | Type: Observational
Why Stopped: CPP requalification
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19-DiVADH; 2019-A00719-48 (Other: IdRCB)
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Hypertensive Disease; Elderly; Vasopressors; General Anesthesia
Keywords: cerebral vasoreactivity; transcranial doppler; hypertensive disease; elderly; vasopressors; general anesthesia
MeSH Terms: conditions — Hypertension | interventions — Ultrasonography, Doppler, Transcranial; Ditiocarb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under vasoconstrictor: Patients older than 65 years old and hypertensive, requiring vasoconstrictor (phenylephrine or Neosynephrine) during general anesthesia.
  Interventions: Other: Transcranial Doppler (DTC)

INTERVENTIONS:
Other: Transcranial Doppler (DTC) — Evaluation of Vasoconstrictor Vasoreactivity with Transcranial Doppler

SUMMARY:
During a general anesthesia, people over 65 years old and hypertensive, have a modification of the vasoreactivity and their cerebral blood flow under vasoconstrictor such as norepinephrine or phenylephrine. We study the variation of the average velocity of the average cerebral artery under vasoconstrictor and during a modification of End Tidal CO2 (EtCO2) by transcranial Doppler.

DETAILED DESCRIPTION:
General anesthesia induces a sympathetic block frequently leading to hypotension, especially in elderly and hypertensive patients. Currently, Phenylephrine (PE) and Norepinephrine (NE) are commonly used in clinical practice to address this arterial pressure drop. Their cardiovascular effects are not exactly the same, even though they both increase mean blood pressure.

Maintenance of mean arterial pressure is not the only hemodynamic goal during general anesthesia in the elderly. Cognitive disorders have been demonstrated during post-anesthetic awakening.

Cerebral hemodynamics is assessed by analyzing the speed of blood flow in the middle cerebral artery using transcranial Doppler (DTC). It measures the systolic and diastolic speed as well as the pulsatility index, which are predictive factors for lowering cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* older over 65 years
* high blood pressure disease
* need general anesthesia
* need vasopressors : norepinephrine or phenylephrine
* temporal window of transcranial doppler is viable

Exclusion Criteria:

* Acute, valvular, rhythmic or ischemic cardiovascular pathology
* severe arthritis (stage 3)
* Intra-cranial pathology
* Significant carotid stenosis (> 40%) or carotid endarterectomy
* Cervical surgery
* Taking a premedication that can modify cerebral vasoreactivity
* Insulin-dependent diabetes for more than 10 years
* Person under judicial protection
* Opposition to data processing

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: population, older over 65 years and hypertensive blood pressure disease with general anesthesia in Tours Hospital in France.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Variation of the velocity of the middle cerebral artery with vasoconstrictors and during a modification of EtCO2. | 48 hours
  Measurements from transcranial doppler velocity of the middle cerebral artery

SECONDARY OUTCOMES:
Variation of cardiac output with vasoconstrictors and during modification of EtCO2. | 48 hours
  Measurements from non invasive device (ClearSight System) of the cardiac output. The ClearSight system quickly connects to the patient by wrapping an inflatable cuff around the finger. Then the system presents cardiac output clearly and simply on the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Marc LAFFON, MD-PhD, Study Director — Univsersity Hospital, Tours